CLINICAL TRIAL: NCT07350967
Title: Magnetic Compression Anastomosis Procedure for Partial Jejuno-ileal Diversion: Evaluating the Feasibility of a Novel Endoscopic Magnetic Metabolic Interventional Therapy
Acronym: 2025/08/EMMIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iIDEAS Group Holdings Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025/08/EMMIT
Record Dates: First submitted 2025-12-26; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Type 2; Bariatric Surgery
Keywords: Magnetic Compression Anastomosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic Compression Anastomosis Procedure for Partial Jejuno-ileal Diversion (Experimental)
  Interventions: Device: Magnetic Compression Anastomosis Procedure for Partial Jejuno-ileal Diversion

INTERVENTIONS:
Device: Magnetic Compression Anastomosis Procedure for Partial Jejuno-ileal Diversion — This is an Investigator Initiated, prospective, single-center, single-arm observational study evaluating feasibility and safety of novel magnetic compression Anastomosis device on the formation of partial jejunoileal diversion among obese patients with Type II Diabetes Mellitus (T2DM). A total of 5 patients will be recruited in the study. Following the administration of general anesthesia, an upper GI endoscope (iIDEAs EMMIT System) with the magnet will be maneuvered to the proximal jejunum. Following this, the snare catheter will release the distal magnet at the designated location, which is approximately 20 cm (± 10 cm) distal to the ligament of Treitz. Concurrently, the lower GI endoscope will be inserted into the terminal ileum through the ileocecal valve. The snare catheter will then assist in positioning the second magnet at the target area, located approximately 20 cm (± 10 cm) proximal to the ileocecal valve. Laparoscopic techniques will be employed

SUMMARY:
English, Hindi and Gujarati

DETAILED DESCRIPTION:
This is an Investigator Initiated, prospective, single-center, single-arm observational study evaluating feasibility and safety of novel magnetic compression Anastomosis device on the formation of partial jejunoileal diversion among obese patients with Type II Diabetes Mellitus (T2DM). A total of 5 patients will be recruited in the study. Following the administration of general anesthesia, an upper GI endoscope (iIDEAs EMMIT System) with the magnet will be maneuvered to the proximal jejunum. Following this, the snare catheter will release the distal magnet at the designated location, which is approximately 20 cm (± 10 cm) distal to the ligament of Treitz. Concurrently, the lower GI endoscope will be inserted into the terminal ileum through the ileocecal valve. The snare catheter will then assist in positioning the second magnet at the target area, located approximately 20 cm (± 10 cm) proximal to the ileocecal valve. Laparoscopic techniques will be employed to maneuver the bowel, aligning the proximal and distal magnets for effective magnetic coupling and observing the ring pair mating via intraoperative imaging (fluoroscopy or plain x-ray). An examination of Duodenum will be conducted for visualization of Duodenal Papilla. The gastroplasty, or other concomitant metabolic surgical procedure, will be conducted in accordance with the standard surgical protocol established by the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are willing and able to give informed consent for participation in the study.
2. Male or Female, aged ≥ 25 years to ≤ 65 years inclusive at the time of informed consent
3. BMI 30-50

   * Prior sleeve gastrectomy (> 12 months) or other metabolic surgical procedures with T2DM (characterized by HbA1c > 6.5%) or weight regain
   * T2DM without a history of gastrectomy or other metabolic surgical procedures (diagnosis for > 6M and <10 yrs) taking at least oral antidiabetic medication with fasting glucose < 200mg/dl and HbA1c >6.5 %
4. Agrees to abstain from any form of additional bariatric or reconstructive surgery that could influence body weight for a duration of 1 year

Exclusion Criteria:

1. Pregnancy or breastfeeding mothers, or individuals planning to become pregnant in next 9-12 months
2. Vulnerable individuals (mentally disabled, physically disabled, prisoner, etc.)
3. Current enrolment in another research study or previous participation within 30 days of enrolment
4. Use of injectable insulin
5. Uncontrolled T2DM
6. Uncontrolled hypertension, dyslipidemia, or sleep apnea
7. Current history of injected Glucagon Like Peptide 1 (GLP1)
8. Evidence of type 1 diabetes or of pancreatic exhaustion, as indicated by a C peptide fasting level less than 1 or, for type 1 diabetes, based on measurable levels of serum anti-GAD-65 autoantibodies or, at investigator's discretion, based on measurable levels of other T1D-associated autoantibodies
9. History of highly unusual or challenging gastrointestinal tract anatomy ascertained through earlier endoscopic examination or other diagnostic imaging
10. Previous intestinal, colonic, or duodenal surgery, excluding bariatric procedures
11. Prior surgical interventions, trauma, prosthetic implants, diseases, or genetic factors that hinder or contraindicate the procedure, including scarring and abnormal anatomical structures
12. History of (or known to be at prohibitive risk for) any of the following diseases of the small bowel or closely related conditions: Crohn's disease or other inflammatory bowel disease, celiac disease, resection for cancer, or intra-abdominal adhesive disease including intussusception, perforated appendix and Meckel's diverticulum
13. Refractory gastroesophageal reflux disease (GERD)
14. Barrett's esophagus
15. Any anatomical anomaly that obstructs orogastric access via gastroscope and catheters, as well as manipulation techniques
16. Presence of an implantable pacemaker or defibrillator
17. Any comorbidity or current physiological condition of the subject that, in the opinion of the surgeon or anesthesiologist, poses safety concerns rendering the subject medically unfit for the procedure. This encompasses any conditions for which endoscopic or laparoscopic surgery would be contraindicated, as well as any significant congenital or acquired anomalies of the gastrointestinal tract at or distal to the magnet placement site

Subjects will be deemed ineligible to participate if they fulfill any of the following criteria:

1. Pregnancy or breastfeeding mothers, or individuals planning to become pregnant in next 9-12 months 2. Vulnerable individuals (mentally disabled, physically disabled, prisoner, etc.) 3. Current enrolment in another research study or previous participation within 30 days of enrolment 4. Use of injectable insulin 5. Uncontrolled T2DM 6. Uncontrolled hypertension, dyslipidemia, or sleep apnea 7. Current history of injected Glucagon Like Peptide 1 (GLP1) 8. Evidence of type 1 diabetes or of pancreatic exhaustion, as indicated by a C peptide fasting level less than 1 or, for type 1 diabetes, based on measurable levels of serum anti-GAD-65 autoantibodies or, at investigator's discretion, based on measurable levels of other T1D-associated autoantibodies 9. History of highly unusual or challenging gastrointestinal tract anatomy ascertained through earlier endoscopic examination or other diagnostic imaging 10. Previous intestinal, colonic, or duodenal surgery, excluding bariatric procedures 11. Prior surgical interventions, trauma, prosthetic implants, diseases, or genetic factors that hinder or contraindicate the procedure, including scarring and abnormal anatomical structures 12. History of (or known to be at prohibitive risk for) any of the following diseases of the small bowel or closely related conditions: Crohn's disease or other inflammatory bowel disease, celiac disease, resection for cancer, or intra-abdominal adhesive disease including intussusception, perforated appendix and Meckel's diverticulum 13. Refractory gastroesophageal reflux disease (GERD) 14. Barrett's esophagus 15. Any anatomical anomaly that obstructs orogastric access via gastroscope and catheters, as well as manipulation techniques 16. Presence of an implantable pacemaker or defibrillator 17. Any comorbidity or current physiological condition of the subject that, in the opinion of the surgeon or anesthesiologist, poses safety concerns rendering the subject medically unfit for the procedure. This encompasses any conditions for which endoscopic or laparoscopic surgery would be contraindicated, as well as any significant congenital or acquired anomalies of the gastrointestinal tract at or distal to the magnet placement site 18. History of small bowel surgery such as small bowel resection 19. Active H. pylori infection (prospective participants with active H. pylori may continue with the screening process if they are treated via medication and re-testing verifies the condition has resolved.) 20. History of chronic or acute pancreatitis 21. Known active hepatitis or active liver disease 22. Symptomatic gallstones or kidney stones or acute cholecystitis 23. History of coagulopathy, upper gastro-intestinal bleeding conditions such as ulcers, gastric varices, strictures, congenital or acquired intestinal telangiectasia 24. Use of anticoagulation therapy (excluding aspirin) which cannot be discontinued for 7 days before and 14 days after the procedure 25. Use of P2Y12 inhibitors (clopidogrel, pasugrel, ticagrelor) which cannot be discontinued for 14 days before and 14 days after the procedure (use of low-dose aspirin allowable) 26. History of serious complications of T2DM including coronary artery disease, hypertension, peripheral vascular disease, diabetic retinopathy, and/or diabetes-related soft tissue infection 27. Taking corticosteroids or drugs known to affect GI motility (e.g. Metoclopramide) 28. Receiving weight loss medications such as Meridia, Xenical, or over-the-counter weight loss medications 29. Persistent anemia, defined as Hgb<10 g dL-1 30. Estimated Glomerular Filtration Rate (eGFR) or Modified of Diet in Renal Disease (MDRD) <30 ml/min/1.73m2 31. Active systemic infection 32. Chemotherapeutic cancer treatment within past 9 months, history of abdominal radiation, or active malignancy within the past 5 years 33. Active illicit substance abuse or alcoholism 34. Unhealed ulcers, bleeding lesions, tumors, or any other lesions at the target site for magnet deployment 35. Anticipated requirement for MR imaging within the first two months following the procedure 36. Any anatomical anomaly that prevents or contraindicates laparoscopic access and general laparoscopic procedures 37. Underwent a surgical or interventional procedure within 30 days prior to the current procedure 38. Any scheduled surgical or interventional procedure planned within 30 days following the current procedure 39. Any stroke or transient ischemic attack (TIA) within six months prior to obtaining consent 40. Any other serological markers likely to be associated with poor outcomes 41. Inability to adhere to the follow-up schedule and assessments 42. Any circumstance that, according to the investigator's judgment, could hinder the completion of follow-up evaluations up to Day 360 (for instance, a health issue that might elevate the risks linked to study involvement or could obstruct the analysis of study findings, failure to comply with the visit timetable, or inadequate adherence to the treatment protocol)

-

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Magnetic Compression Anastomosis Procedure for Partial Jejuno-ileal Diversion: Evaluating the Feasibility of a Novel Endoscopic Magnetic Metabolic Interventional Therapy | 1 year
  To evaluate feasibility of the magnetic compression anastomosis system in the development of partial jejunoileal diversion measured by evaluating Magnet placement success rate Passage of magnets without surgical re-intervention Radiological confirmation of patent anastomosis Primary feasibility endpoints will be met if the device performance is confirmed in more than 80 percent of treated safety

CONTACTS AND LOCATIONS:
Locations (1):
- AB Plus Speciality Hospital, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No